CLINICAL TRIAL: NCT01847066
Title: Fractional Erbium 2940nm Laser & Impact US for Trans-Epidermal Delivery of Cosmetic Anti-Aging Ingredients for Wrinkles, Acne Scars and Pigmented Skin: A Randomized Split Face & Dorsal Hand Side by Side Study
Brief Title: Epidermal Delivery of Ani-Aging Ingredients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Alma Lasers Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALMA 013-001
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Wrinkles; Acne Scars; Pigmentation
Keywords: wrinkles; acne scars; pigmentation
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Erbium plus cosmetics plus Impact (Active Comparator): Erbium 2940 plus cosmetics plus Impact Patient shall be treated with erbium 2940nm laser, cosmetics and the Impact.
  Interventions: Device: Erbium 2940 plus cosmetics plus Impact
- Erbium 2940 plus cosmetics (Active Comparator): Erbium 2940 plus cosmetics Patient shall be treated with erbium 2940nm laser, cosmetics
  Interventions: Device: Erbium 2940 plus cosmetics
- Erbium 2940 plus cosmetics plus Impact (Active Comparator): Patient shall be treated with erbium 2940nm laser, cosmetics and the Impact.
  Interventions: Device: Erbium 2940 plus cosmetics plus Impact
- Erbium 2940nm plus cosmetics (Active Comparator): Patients shall be treated with Erbium 2940nm laser plus cosmetics only.
  Interventions: Device: Erbium 2940 plus cosmetics

INTERVENTIONS:
Device: Erbium 2940 plus cosmetics plus Impact — Laser used in all arms
  Other Names: Laser
  Arms: Erbium 2940 plus cosmetics plus Impact; Erbium plus cosmetics plus Impact
Device: Erbium 2940 plus cosmetics — laser
  Other Names: Laser
  Arms: Erbium 2940 plus cosmetics; Erbium 2940nm plus cosmetics

SUMMARY:
To assess the safety and efficacy of an ablative fractional, 2940-nm laser combined with the US Impact and cosmetic -formulations for improving the appearance of wrinkles, acne scars and pigmented skin.

DETAILED DESCRIPTION:
This is a randomized, split face & dorsal hand side by side study. The purpose of the side by side study is to determine whether the use of the Impact with the ablative fractional 2940nm laser and cosmetics improves the cosmetic outcomes when compared to using just the ablative fractional 2940nm laser with the cosmetics.

This is a non-significant risk aesthetic clinical study. Only cosmetic formulations will be used during the study, These cosmetic formulations do not contain any ingredient categorized as a drug by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female in good general health between 35 to 65 years of age.
* Must be willing to execute informed consent. Patient must also consent to having photos taken at each visit.
* A potential subject must exhibit:

Facial wrinkling, acne scars or pigmentation.

* For FEMALE PATIENTS OF CHILDBEARING POTENTIAL, must have had a regular menstrual cycle prior to study entry (a female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation) and is willing to use an acceptable form of birth control during the entire course of the study [i.e., acceptable methods of birth control are oral contraceptives, contraceptive patches/rings/implants Norplanit®, Depo-Provena®, double-barrier methods (e.g. condoms and spermicide), abstinence and vasectomies of partner with a documented second acceptable method of birth control should the subject become sexually active]. All systemic birth control measures must be in consistent use at least 30 days prior to study participation.
* Must be willing to comply with study visits and complete the entire course of the study.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from participation:

The following are exclusion criteria for subjects in this study:

* A subject that underwent a laser / light treatment on the face within 12 months, or any topical treatment on the face with 6 months.
* A subject with any UNCONTROLLED systemic disease. A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
* A subject with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
* A subject using any topical product containing a retinoid, retinol, or other vitamin A derivative within 3 months prior to or during the study period.
* A subject using any systemic steroid therapy within 6 months prior to or during the study period.
* A subject that has been treated with Botox/Dysport or filler/biostimulatory molecule injections to his/her face within the past six months.
* A subject using any topical medicated creams, lotions, powders, etc. on the treatment areas during the study period, other than the study treatment regimen within 14 days.
* A subject that has previously been treated with systemic retinoids within the past year (e.g., Accutane®, Roche Dermatologics).
* A subject with recently excessive facial exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing). During the study, when excessive sun exposure is unavoidable, subjects must wear appropriate protective clothing (e.g. hat) and comply with the study dosing regimen of daily application of the dispersed sunblock.
* A subject with a recent history or active presence of any facial skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e. moderate to severe acne vulgaris, atopic dermatitis, psoriasis, rosacea, seborrheic dermatitis, excessive facial hair or coloration).
* A female subject who is pregnant, nursing an infant or planning a pregnancy during the study [throughout the course of the study, women of child-bearing potential must use reliable forms of contraception (i.e., oral contraceptive, intrauterine device, abstinence, or spermicides and condoms used in combination)].
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.
* Subjects who are pregnant, breast-feeding, or planning a pregnancy. Females of childbearing potential, must be either:
* using the same form (i.e. brand) and dosage regimen of an oral contraceptive pill or of a hormonal implant continuously for three months prior to study entry and continue during the entire study, or
* willing to use a different form of birth control during the study other than any form of hormonal methods such as oral contraceptive pills and hormonal implants 30 day prior to study entry and during the entire study period. For the purpose of this study, the following are considered acceptable methods of birth control: double-barrier methods (e.g.: condoms and spermicide), abstinence and vasectomies of partner with a documented second acceptable method of birth control should the subject become sexually active.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Photographs to determine improvement of appearance | 4 months
  An independent panel of qualified blinded physicians (masked) with respect to subject-identity, photo chronology, treatment methodology (with/without Impact module), study time point, and treatment assignment will grade the photographs as determined by:
  1. Clinical Photographs Alexiades-Armenakas Grading Scale Assessment
  2. Clinical Photographs Acne Scar Grading Scale (see section 7.1)
  3. Clinical Photographs Hand Pigmentation Grading Scale (see section 7.1)
  4. Spectrophotometric (Reflectance Spectroscopy) Analysis of La*b* values

CONTACTS AND LOCATIONS:
Locations (1):
- NY Derm LLC, New York, New York, United States